CLINICAL TRIAL: NCT06964646
Title: Efficacy, Safety, and Tolerability of 8 Weeks of Vaginal Hyaluronic (V-HYAL) Gel in Peri- and Post-Menopausal Female
Brief Title: Assess Efficacy, Safety, and Tolerability of 8 Weeks of Vaginal Hyaluronic (V-HYAL) Gel in Peri- and Post-Menopausal Female
Acronym: V-HYAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VDMEN-V4.0-2023; NMRR ID-23-02085-IH7 (Other: National Institute of Health Malaysia)
Record Dates: First submitted 2025-04-09; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Vaginal Dryness

STUDY DESIGN:
Intervention Model Description: The intervention group received repeat doses of 2.5g of V-HYAL Gel® (formerly Vaginal Hyal Gel) every three days, while the control group did not receive the gel.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (with V-HYAL Gel (formerly Vaginal Hyal Gel)) (Experimental): Given 2.5g of Vaginal Hyal gel
  Interventions: Drug: Vaginal Hyal gel 2.5g
- Control group (No Intervention): No intervention control group

INTERVENTIONS:
Drug: Vaginal Hyal gel 2.5g — vaginal gel 2.5g
  Arms: Intervention Group (with V-HYAL Gel (formerly Vaginal Hyal Gel))

SUMMARY:
The goal of this clinical trial is to assess the efficacy of repeat doses of V-HYAL Gel on vaginal dryness in Peri- and Post-Menopausal Female. The main questions it aims to answer :

* To evaluate the effect of V-HYAL Gel on subjects' quality life.
* To evaluate the effect of V-HYAL Gel on the vaginal lactobacillus flora, vaginal thrush, bacterial vaginosis and trichomonas vaginalis
* To evaluate the safety and tolerability of repeat doses of V-HYAL Gel. Researchers will compare V-Hyal treated arm to see for its efficacy and safety.

Participants will have screening visit for the evaluation of subject's eligibility and three study days, Day 0 (Baseline), Week 4 (Telephone contact), and Week 8 (End of study visit). Primary criterion: Visual Analogic Scale (VAS) of vaginal dryness Secondary criterion: Vaginal microbiota and immunology HRQoL(SF 8), DIVA, FSFI questionnaires Patient Global Impression of Improvement Vaginal PH VHI scale.

DETAILED DESCRIPTION:
Primary outcome:

The primary outcome was the subjective performance evaluation in terms of the Visual Analogic Scale (VAS) for vaginal dryness was used as the primary criteria for determining the results of the trial. VAS was assessed at baseline (Day 0), during a telephone contact after the fifth administration, and at the final visit (week 8) after 19 administrations. VAS assessed are vaginal dryness, vaginal itching, vaginal irritation, and painful urination (0-10, 0 = absent, 10 = intolerable). Between-group differences in the proportion of patients with a reduction in VAS score at week 8, at p-value < 0.05 significant.

Secondary outcome:

Criteria to be used as secondary outcomes are as follows:

* High vaginal swab (HVS) to measure vagina lactobacillus flora, vaginal thrush, bacterial vaginosis and trichomonas vaginalis was done by taking a High Vaginal Swab (HVS) from the posterior fornix and observing the intensity and variety of microflora.
* pH measurements were taken using pH strips.
* Adverse events include any form of vaginal bleeding, bothersome vaginal irritations, bacterial vaginosis, vaginal yeast infection and hypersensitivity reactions.
* Vaginal Health Index (VHI) (cut-off < 15 index of atrophic vagina) and between-group difference in mean change from baseline to end of study (week 8) Female Sexual Function Index Scoring (FSFI)
* Day-to-day Impact of Vaginal Aging Questionnaire (DIVA)

ELIGIBILITY:
Inclusion Criteria:

1. Peri or post-menopausal.
2. BMI between 18 kg/m2 and 30 kg/m2.
3. Able to give written informed consent before starting any study-related procedure.
4. Medical history and physical examination normal or abnormal but not clinically relevant on the investigator judgment.
5. ECG tracing, blood pressure and laboratory tests within normal range or abnormal but not clinically relevant as per the investigator's judgment.
6. Not under any administrative or legal supervision.
7. Sexually active in the last three months

Exclusion Criteria:

1. Inability or unwillingness to comply with the requirements of the protocol as determined by the investigator.
2. Inability or unwillingness to provide written consent.
3. Pregnancy, breastfeeding, or use of nonreliable methods of contraception.
4. Other medical conditions which, in the investigator's judgment, may be associated with increased risk to the subject or may interfere with study assessments or outcomes.
5. History or evidence of allergy, idiosyncrasy or hypersensitivity to hyaluronic acid.
6. History or clinical evidence of significant or uncontrolled cardiovascular, respiratory, renal, hepatic, endocrine, metabolic, gastrointestinal, haematological, neurological or psychiatric pathology which may affect the study outcomes.
7. Chronic diseases such as HIV I and II, HBV and HCV surgery within previous 6 months, or blood loss > 400 mL within previous 3 months.
8. History of alcohol or drug abuse.
9. Took hormone therapy or tibolone in the 3 months before the first dosing occasion and during the study.
10. Took any pharmacological treatment which may affect the vaginal dryness or study outcomes, such as Menopausal Hormone Therapy (except for symptomatic short-term paracetamol use)
11. Received concomitant treatment with other investigational drugs or had participated in another clinical trial within the previous 6 months prior to dosing / 4 weeks prior to screening visit.
12. Had any surgery or medical treatment which may interfere with study outcomes (i.e. hysterectomy).
13. Any subject who cannot be contacted in case of emergency.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is specific to the biological female sex as it involves female reproductive organ
Enrollment: 70 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Visual Analogic Scale (VAS) | . VAS was assessed at baseline (Day 0), during a telephone contact after the fifth administration (Week 4), and at the final visit (week 8) after 19 administrations.
  Subjective performance evaluation in terms of the Visual Analogic Scale (VAS) for vaginal dryness was used as the primary criteria for determining the results of the trial.VAS assessed are vaginal dryness, vaginal itching, vaginal irritation, and painful urination (0-10, 0 = absent, 10 = intolerable). Between-group differences in the proportion of patients with a reduction in VAS score at week 8, at p-value < 0.05 significant.

SECONDARY OUTCOMES:
High Vaginal Swab | 8 weeks
  Measure vagina lactobacillus flora, vaginal thrush, bacterial vaginosis and trichomonas vaginalis was done by taking a High Vaginal Swab (HVS) from the posterior fornix and observing the intensity and variety of microflora
Vaginal pH | 8 weeks
  pH measurements were taken using pH strips before and after using the investigational product
Vaginal Health Index | 8 weeks
  Vaginal Health Index (VHI) (cut-off < 15 index of atrophic vagina) and between-group difference in mean change from baseline to end of study (week 8)
Female Sexual Function Index Scoring (FSFI) | 8 weeks
  Female Sexual Function Index Scoring (FSFI) between-group difference in mean change from baseline to end of study (week 8) The Female Sexual Function Index (FSFI) is a standardized, 19-item questionnaire used to assess sexual function in women across six key domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Each domain includes a specific number of questions with responses scored on a Likert scale, typically ranging from 0 or 1 to 5. Domain scores are calculated by summing the scores of the relevant questions and multiplying by a domain-specific factor: desire (×0.6), arousal (×0.3), lubrication (×0.3), orgasm (×0.4), satisfaction (×0.4), and pain (×0.4). The total FSFI score is the sum of these six domain scores, with a maximum possible score of 36. A total score of 26.55 or lower is generally considered indicative of female sexual dysfunction.
Day-to-day Impact of Vaginal Aging (DIVA) | 8 weeks
  The DIVA questionnaire includes 23 items distributed across four domains: daily activities (5 items), emotional well-being (4 items), sexual functioning (9 items), and self-concept/body image (5 items). Each item is rated on a 5-point Likert scale from 1 (no impact) to 5 (very severe impact), with higher scores indicating greater negative impact. For each domain, the scores of individual items are averaged to produce a mean domain score, rather than summed, ensuring comparability across domains with different numbers of items.

CONTACTS AND LOCATIONS:
Overall Officials: Hasniza Zaman Huri Prof, Doctor of Philosophy, Study Chair — University of Malaya
Locations (1):
- Hospital Seberang Jaya, Seberang Jaya, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen J, Geng L, Song X, Li H, Giordan N, Liao Q. Evaluation of the efficacy and safety of hyaluronic acid vaginal gel to ease vaginal dryness: a multicenter, randomized, controlled, open-label, parallel-group, clinical trial. J Sex Med. 2013 Jun;10(6):1575-84. doi: 10.1111/jsm.12125. Epub 2013 Apr 9. PMID 23574713